CLINICAL TRIAL: NCT02020109
Title: Evaluation of Splenic Irradiation in Chronic Lymphatic Leukemia (CLL)
Brief Title: Evaluation of Splenic Irradiation in Chronic Lymphatic Leukemia
Status: Withdrawn | Type: Observational
Why Stopped: Logistics and financial
Sponsor: Maastricht Radiation Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: 13-11-05/06-extern-6295
Record Dates: First submitted 2013-12-12; First posted 2013-12-24 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Leukemia, Chronic Lymphatic
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with Chronic Lymphatic Leukemia: Patients with Chronic Lymphatic Leukemia treated with splenic irradiation
  Interventions: Radiation: splenic irradiation

INTERVENTIONS:
Radiation: splenic irradiation

SUMMARY:
Retrospective evaluation on the effect of splenic irradiation on clinical and hematological response and toxicity in patients with chronic lymphatic leukaemia (CLL).

DETAILED DESCRIPTION:
The study will include patients with CLL treated with splenic irradiation in Maastro Clinic, Maastricht, The Netherlands, Maxima Medisch Centrum Veldhoven/Catharina hospital, Eindhoven, The Netherlands and Modena hospital, Modena, Italy. Data will be collected from patient records in an uniform database. Data will include demographic data, CLL stadium (RAI and Binet) at diagnosis and at the time of irradiation treatment, clinical data at diagnosis (haematology), splenic irradiation data, follow-up data such as date of progression or death

ELIGIBILITY:
Inclusion Criteria:

* patients with chronic lymphatic leukaemia.

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic lymphatic leukaemia (CLL).
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-09; Primary Completion 2016-12 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Clinical and haematological response | 13 years
  Clinical and haematological response measured by number of leucocytes and thrombocytes during and after irradiation. Hemoglobin and size of spleen during and after irradiation in the time period 2000 tot 2013

SECONDARY OUTCOMES:
Progression of chronic Lymphatic leukaemia | 13 years
  Progression of chronic Lymphatic leukaemia after irradiation in the time period 2000 tot 2013
Death | 13 years
  Patients will be followed from the time of splenic irradiation to death in the time period of 2000 tot 2013
Toxicity of splenic irradiation | 13 years
  Toxicity of splenic irradiation during and after irradiation measured by evaluating clinical toxicity based on the CTCAE version 3.0 during and after irradiation (2000 to 2013)

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Borger, dr., Principal Investigator — Maastro Clinic, The Netherlands
Locations (1):
- Maastro Clinic, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided